CLINICAL TRIAL: NCT05095038
Title: A Six Month Randomized Placebo-controlled Trial of Appethyl® vs Placebo in Management of Pre-diabetes on Overweight and Obese Individuals
Brief Title: The Effect of Appethyl® vs Placebo on Human Health (Appethyl)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The collaborator providing funding for the study has suspended the payment
Sponsor: University of Copenhagen (Other)
Collaborators: Greenleaf Medical AB, Lund, Sweden (Unknown); Lund University (Other)
Responsible Party: Principal Investigator, Faidon Magkos, Principal Investigator, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: B368; H-21045373 (Registry Identifier: Danish Ethical Committee)
Record Dates: First submitted 2021-09-22; First posted 2021-10-27 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Overweight and Obesity; PreDiabetes
Keywords: Appetite; Bodyweight; Fasting blood glucose; Blood lipids; Body composition
MeSH Terms: conditions — Overweight; Obesity; Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Appethyl® (Experimental): Participants are instructed to ingest 10 capsules daily and they are instructed to swallow the capsules in whole with a glass of water with/during lunchtime throughout the study period of 26 weeks.
  Each capsule contain 0.5 g Appethyl®, and the daily intake is 5 g/day.
  Interventions: Dietary Supplement: Appethyl®
- Placebo (Placebo Comparator): Participants are instructed to ingest 10 capsules daily and they are instructed to swallow the capsules in whole with a glass of water with/during lunchtime throughout the study period of 26 weeks.
  Each capsule contain 0.5 g placebo, and the daily intake is 5 g/day.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Appethyl® — Spinach extract, capsules, 5g/day, 26 weeks.
  Arms: Appethyl®
Dietary Supplement: Placebo — Pea protein, capsules, 5g/day, 26 weeks.
  Arms: Placebo

SUMMARY:
The study will be conducted as a 26-week double-blinded randomized placebo-controlled trial of Appethyl® vs placebo in 100 overweight/obese (BMI ≥25.0-35.9 kg/m^2) men and women between 18-65 years with prediabetes (fasting plasma glucose of 5.6 mmol/L to <7.0 mmol/L). At initiation, all subjects will receive healthy life style instructions in accordance to the guidelines described in the Nordic Nutrition Recommendations.

The study aim to investigate the effect over time (26-weeks) of daily Appethyl® treatment compared to placebo on change in fasting glucose (primary endpoint) and several other health markers (secondary endpoint).

The hypothesis to be tested is whether the null hypothesis (no difference between Appethyl® and placebo with regard to endpoint data) can be rejected.

ELIGIBILITY:
Inclusion Criteria:

* Male and women Age between 18-65 years
* BMI ≥25.0-35.9 kg/m^2
* Prediabetes (defined according to ADA with a fasting plasma glucose of 5.6 mmol/L to <7.0 mmol/L)
* Provided voluntary written informed consent

Exclusion Criteria:

* Non-covid-19 vaccinated
* Known diseases which may affect energy expenditure and/or satiation/satiety/food intake
* History or diagnosis of eating disorder
* Any physical abnormality or medical condition which might have impact on following the dietary regimen
* Psychiatric disorders i.e. schizophrenia, bipolar disease or depression with hospitalization within the last 6 months
* Diabetes mellitus (type 1 and 2)
* History or diagnosis of cardiovascular disease, chronic kidney disease, liver disease and cancer
* Known systolic blood pressure above 160 mmHg and/or diastolic blood pressure above 100 mmHg whether on or off treatment for hypertension. If being treated, stable treatment (i.e. no change in treatment, either dose, type of medication or other changes) within last three months is required
* Active inflammatory bowel disease, celiac disease, chronic pancreatitis or other disorder potentially causing malabsorption
* Systemic treatment with glucocorticoids inhalations and creams etc. is allowed
* Previous bariatric surgery or intention to undergo bariatric surgery within the next 12 months
* History of extensive small or large bowel resection
* Known endocrine origin of obesity (except for treated hypothyroidism)
* Transmissible blood-borne diseases e.g. hepatitis B, HIV
* Any recent surgical procedure not fully recovered (as judged by the investigator)
* Current use of prescription medication or use within the previous month that has the potential of affecting body weight
* Current use of other prescription medication that does not affect body weight should have been stable for the past three months and expected to be stable during the study
* Concurrent therapy with immunosuppressive drugs or cytotoxic agents
* Hemoglobin concentration below local laboratory reference values (i.e. anemia)
* Being lactating, pregnant or planning to become pregnant within the study period
* Weight changes ± 5% three months prior inclusion
* Dietary patterns interfering with the study protocol, as judged by the investigator, two months prior inclusion, during the study or plans to initiate during the study
* Use of pre- and probiotic products (incl. fiber supplements) within one month prior to study initiation as well as during the study (except psyllium 10 g/day)
* Use of dietary supplementation should be stable three months prior to study initiation as well as during the study
* Severe food allergies and food intolerances expected to interfere with the study
* Intolerance, allergy or dislike of intervention products (e.g. pea allergy)
* Engagement in elite sports or similar strenuous exercise ≥5 h/week
* Blood donation or transfusion within the past month before screening
* Planned blood donation for other purpose than this study during participation
* Consumption of alcohol corresponding to >2 (for men) and >1 (for women) units/day
* Drug abuse, as judged by the investigator, within the previous 12 months
* Psychological or behavioral problems which, in the judgement of the investigator, would lead to difficulty in complying with the study protocol
* Participation in other clinical trials within the past three months or intention to do so during the study, which are likely to affect the present study
* Unable to consume the interventional product for religious reasons, swallowing disorders, other physiological reasons or any other reasons for not being able to follow the recommended diet
* Inability or unwillingness to give written informed consent or communicate with study personnel
* Inability or unwillingness to follow the study protocol and instructions given by the study personnel
* Illiteracy or inadequate understanding of Danish/Scandinavia
* Any other condition that judged by the investigator may interfere with the adherence to the study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Fasting blood glucose | Change from baseline (week 0) to end of intervention (week 26)
  To investigate the effect over time of daily Appethyl® treatment compared to placebo on change in fasting glucose.

SECONDARY OUTCOMES:
Change in bodyweight | Change from baseline (week 0) to end of intervention (week 26)
  Body weight will be measured at baseline (week 0), week 12 and after end of intervention (week 26) in a fasting state. Body weight will be measured wearing only underwear or light clothing as well as no shoes and stockings. Body weight will be measured on a calibrated scale and subjects will be instructed to stand in the middle of the platform of the scale with straight neck and eyes looking straight ahead, whilst distributing their weight evenly on body feet after having emptied their bladder. Two measurements are made when the scale has stabilized and both results are recorded to the nearest 0.1 kg and the average of the two measurements is used for further analysis.
Change in fasting Insulin | Change from baseline (week 0) to end of intervention (week 26)
  Venous blood samples will be collected at baseline (week 0), week 12 and after end of intervention (week 26) by a vein puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. HOMA-IR and HOMA-IS will be calculated from fasting blood glucose and insulin concentrations.
Change in hbA1c | Change from baseline (week 0) to end of intervention (week 26)
  Venous blood samples will be collected at baseline (week 0), week 12 and after end of intervention (week 26) by a vein puncture in the antecubital vein after an overnight fast from at least 10 pm the night before.
Change in anthropometrics | Change from baseline (week 0) to end of intervention (week 26)
  Waist- and hip circumference will be measured at baseline (week 0), week 12 and after end of intervention (week 26) in a fasting state. The measurements of waist- and hip circumference will be performed with an empty bladder and performed with a non-elastic tape measuring. Waist circumference is measured mid-way between the lower rib and iliac crest (top of the hip bone) at the end of expiration with the subject in a standing position with their weight distributed evenly on both feet. Hip circumference is measures at the widest point between the hips and buttocks observed from the front at the end of expiration with the subject in a standing position with their weight distributed evenly on both feet. Two measurements of waist- and hip circumference will be made and both results will be recorded to the nearest 0.5 cm and the average of the two measurements is used in further analysis
Change in body composition | Change from baseline (week 0) to end of intervention (week 26)
  Body composition will be assessed by a whole body DXA scan at baseline (week 0), week 12 and after end of intervention (week 26) assessing lean mass (kg), fat mass (kg), abdominal fat (kg), visceral fat (kg) and bone mineral density (g/cm^2). The DXA scan will be performed in a fasting condition with the subjects only wearing light clothing and after emptying the bladder.
Change in inflammation | Change from baseline (week 0) to end of intervention (week 26)
  Venous blood samples will be collected at baseline (week 0), week 12 and after end of intervention (week 26) by a vein puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Leptin (pg/ml), adiponectin (ng/ml), IL-6 (pg/ml), TNF-alfa (pg/ml) and hsCRP (mg/L) will be assessed.
Change in blood lipids | Change from baseline (week 0) to end of intervention (week 26)
  Venous blood samples will be collected at baseline (week 0), week 12 and after end of intervention (week 26) by a vein puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Blood lipids: LDL and TG
Change in blood pressure | Change from baseline (week 0) to end of intervention (week 26)
  Systolic and diastolic blood pressure (mmHg) will be measured at baseline (week 0), week 12 and after end of intervention (week 26) using a validated automatic device. The blood pressure will be measured on the right arm with an appropriate arm cuff after 5-10 min rest in a resting position. The measurement will be performed three times approximately two minutes apart, and the reading is recorded to the nearest 1 mmHg for blood pressure. A mean value of the three readings will be used in further analysis.
Change in pulse | Change from baseline (week 0) to end of intervention (week 26)
  Pulse (beats per minute) will be measured at baseline (week 0), week 12 and after end of intervention (week 26) using a validated automatic device. The pulse will be measured on the right arm with an appropriate arm cuff after 5-10 min rest in a resting position. The measurement will be performed three times approximately two minutes apart, and the reading is recorded to the nearest 1 beats per minute for pulse. A mean value of the three readings will be used in further analysis.
Change in the proportion of participants converting to normoglycemia | Change from baseline (week 0) to end of intervention (week 26)
  Number of participants converting from prediabetes to normal glucose levels
Change in subjective assessment of dietary preferences | Change from baseline (week 0) to end of intervention (week 26)
  Subjective measurements of hunger, satiety, taste for sweet, fat and salt will be assessed by Visual Analogue Scales (VAS) (0-10 cm, where 10 being the highest ranking). The participants will be asked to complete the VAS at baseline (week 0) and at every visit from week 0 to 26 (week 4, 8, 12, 16, 20 and 24). Moreover, every fourth week from week 2 to week 22 (week 2, 6, 10, 14, 18, and 22) participants will be asked to complete the questionnaire regarding subjective assessment of dietary preferences at home. The questionnaire will be handed out prior to completion.
Change in subjective assessment of investigational product | Change from baseline (week 0) to end of intervention (week 26)
  Participants will be asked to answer a questionnaire (on a scale from 1-5 going from very tolerable to very intolerable) regarding their experience of the investigational product at baseline (week 0) and at every visit from week 0 to 26 (week 4, 8, 12, 16, 20 and 24). Moreover, every fourth week from week 2 to 22 (week 2, 6, 10, 14, 18, and 22) participants will be asked to complete the questionnaire regarding subjective assessment of the investigational product at home. The questionnaire will be handed out prior to completion.

CONTACTS AND LOCATIONS:
Overall Officials: Faidon Magkos, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Frederiksberg, DK, Denmark

IPD SHARING:
Plan to Share IPD: No